CLINICAL TRIAL: NCT05580263
Title: The Effect of Different Order of Concurrent Training Consisting Aerobic and Resistance Exercise on Improving Visceral Adipose Tissue and Insulin Resistance for Community Residents With Obesity.
Brief Title: Different Order of Concurrent Training on Improving Visceral Adipose Tissue and Insulin Resistance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Tainan Junior College of Nursing (Other)
Responsible Party: Principal Investigator, Yu-Hsuan Chang, Assistant professor, National Tainan Junior College of Nursing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 110-551
Record Dates: First submitted 2022-10-03; First posted 2022-10-14 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Fat Burn; Aerobic Exercise; Resistance Exercise
MeSH Terms: interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: PI (data assessor) will be blinded for the grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aerobic exercise(AE) preceding resistance exercise(RE) (Experimental): at least moderate intensity of AE 30 minutes than RE 15 minutes, with a break of 5 minutes between two modalities of training.
  Interventions: Behavioral: aerobic exercise; Behavioral: resistance exercise
- RE preceding AE (Experimental): RE 15 minutes than at least moderate intensity of AE 30 minutes, with a break of 5 minutes between two modalities of training.
  Interventions: Behavioral: aerobic exercise; Behavioral: resistance exercise
- Control group (No Intervention): Participants maintain their usual life without any exercise intervention.

INTERVENTIONS:
Behavioral: aerobic exercise — The main AE program will be designed and controlled for at least moderate intensity of heart rate reserve (HRR) lasting 30 minutes. The goal of intensity will be set at least 40% of HRR during the first two weeks, and then progressively increase the targeted intensity at the end of 16 weeks with 60% HRR. The motions will design by involving core muscle training (e.g., march, step touch, lunge, V-step, box step, twist, knee up, scoop, and scissors).
  Arms: RE preceding AE; aerobic exercise(AE) preceding resistance exercise(RE)
Behavioral: resistance exercise — In the process, the participants will be instructed by resisting the weight smoothly, and peaking at hold. RE prescription consist of 2-4 sets with 10-15 repetitions per set with a rest interval of 1-2 minutes between sets to improve muscular fitness.
  The first two weeks will start with two sets of 10-15 repetitions and then gradually progress on four sets of 15 repetitions at the end of 16 weeks. The total duration of RE will lasting around 15 minutes.
  Arms: RE preceding AE; aerobic exercise(AE) preceding resistance exercise(RE)

SUMMARY:
Purposes: The purpose of one-year project is to compare the effect of different intrasession exercise order of AE and RE during concurrent training on reducing VAT and improving insulin resistance for inactive middle-age community residents with obesity.

Methods: Purposive sampling will be used to enroll community residents aged 40-64 years with inactive habit and body fat percentage ≧ 25% for male and ≧ 30% for female in southern Taiwan. Eligible participants will be stratified by sex and age (40-55years and 56-64 years) then block randomly divided into training group of AE preceding RE, RE preceding AE or a control group. The exercise training program will under supervision lasting 16 weeks with 3 times per week. The concurrent training prescription consist of AE 30 minutes and RE 15 minutes per session. A 5-minute interval between two exercise modalities. All participants will be evaluated outcomes for two time points including baseline (T0) and after 16-week intervention (T1). The primary outcomes are VAT and insulin resistance. A two-way ANOVA with repeated measures will be performed to compare changes of outcome variables over the intervention period.

Relevance to clinical practice: The results of this project can assist health professionals to know how to properly prescribe concurrent training of AE and RE to achieve the greatest effects on VATreduction and insulin resistance improvement for middle-age residents with obesity.

DETAILED DESCRIPTION:
Background: Visceral adipose tissue (VAT) accumulation is highly linking with cardiovascular diseases and insulin resistance. A combination of aerobic exercise (AE) and resistance exercise (RE) was an effective strategy to improve VAT and insulin resistance; however, no current evidence displayed whether the different orders of concurrent training (AE preceding RE or RE preceding AE) influence the effects on VAT reduction and insulin resistance improvement.

Purposes: The purpose of one-year project is to compare the effect of different intrasession exercise order of AE and RE during concurrent training on reducing VAT and improving insulin resistance for inactive middle-age community residents with obesity.

Methods: Purposive sampling will be used to enroll community residents aged 40-64 years with inactive habit and body fat percentage ≧ 25% for male and ≧ 30% for female in Tainan. Eligible participants will be stratified by sex and age (40-55years and 56-64 years) then block randomly divided into training group of AE preceding RE, RE preceding AE or a control group. The exercise training program will under supervision lasting 16 weeks with 3 times per week. The concurrent training prescription consist of AE 30 minutes and RE 15 minutes per session. A 5-minute interval between two exercise modalities. The control group will follow their primary lifestyle without exercise intervention. All participants will be evaluated outcomes for two time points including baseline (T0) and after 16-week intervention (T1). The primary outcomes are VAT and insulin resistance. VAT is measured by body composition analyzer and insulin resistance is calculate from fasting glucose and insulin level in blood samples. A two-way ANOVA with repeated measures will be performed to compare changes of outcome variables over the intervention period.

Relevance to clinical practice: The results of this project can assist health professionals to know how to properly prescribe concurrent training of AE and RE to achieve the greatest effects on VATreduction and insulin resistance improvement for middle-age residents with obesity.

ELIGIBILITY:
Inclusion Criteria:

* 40 to 64 years old.
* body fat percentage ≧ 25% for male and ≧ 30% for female.
* with inactive habit (≤ 3 days of physical activity per week and ≤ 30 min per session).
* can communicate in Mandarin or Taiwanese.

Exclusion Criteria:

* with recent unstable conditions in which had potential risk on exercise including stroke, cardiovascular and respiratory diseases, handicap, pregnancy.
* with any contraindications to body composition analyzer measurement including body embed pacemakers and artificial metal joints, amputated hands or feet.
* cannot corporate with either examination or intervention.
* use psychotropic or appetite-regulating medicine.
* under oral hopoglycemic agent or insulin treatment.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
visceral adipose tissue | at baseline
  Participants will measure visceral adipose tissue measure at baseline by body composition analyzer.
visceral adipose tissue | 16-week after intervention
  Participants will measure visceral adipose tissue measure after 16-week intervention by body composition analyzer.
Insulin | at baseline
  Participants will collect insulin at baseline by blood samples
Insulin | 16-week after intervention
  Participants will collect insulin after 16-week intervention by blood samples
Fasting glucose | at baseline
  Participants will collect fasting glucose at baseline by blood samples
Fasting glucose | 16-week after intervention
  Participants will collect fasting glucose after 16-week intervention by blood samples

SECONDARY OUTCOMES:
waist circumference | at baseline
  Participants will measure waist circumference at baseline by tape measurement
waist circumference | 16-week after intervention
  Participants will measure waist circumference after 16-week intervention by tape measurement
hip circumference | at baseline
  Participants will measure hip circumference at baseline by tape measurement
hip circumference | 16-week after intervention
  Participants will measure hip circumference after 16-week intervention by tape measurement
weight | at baseline
  Participants will measure weight at baseline by body composition analyzer
weight | 16-week after intervention
  Participants will measure weight after 16-week intervention by body composition analyzer
body fat percentage | at baseline
  Participants will measure body fat percentage at baseline by body composition analyzer
body fat percentage | 16-week after intervention
  Participants will measure body fat percentage after 16-week intervention by body composition analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsuan Chang, phD, Principal Investigator — National Tainan Junior College of Nursing
Locations (1):
- Natioal Tainan Junior College of Nursing, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data available on request due to privacy/ethical restrictions